CLINICAL TRIAL: NCT00001523
Title: Structure and Functional Status of Parotid Glands Exposed to Therapeutic Irradiation
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960082; 96-D-0082
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Radiation Injuries; Xerostomia
Keywords: Cytology; Diagnostic Imaging; Radiation Damage; Saliva; Serostomia; Xerostomia; Head Cancer; Neck Cancer
MeSH Terms: conditions — Radiation Injuries; Xerostomia; Head and Neck Neoplasms

SUMMARY:
Therapeutic irradiation to the head and neck for cancer damages salivary glands present in the radiation field. Despite long recognition of radiation-induced salivary hypofunction, and the associated oral morbidities, the specific damage mechanism(s) is not known and the structure and functional integrity of the surviving parenchymal tissue has not been well-documented. Detailed knowledge of the latter is particularly necessary in order to design appropriate corrective therapies. It is the purpose of this study to provide such a detailed structural and functional assessment of human parotid glands following irradiation. The study will examine 20 patients beginning just prior to therapeutic irradiation and continuing at intervals for 3 years for a total of 5 study visits. Study visits (prior to irradiation and at 4 weeks, 12 weeks, 12 months and 36 months post-irradiation) will include the following procedures: i) detailed oral exam and structured interview; ii) salivary gland functional assessment; iii) sialography of each parotid gland; iv) 99mTcO4 scan of the salivary glands; and v) a magnetic resonance imaging (MRI) scan of the parotid glands. Based on previous single observation studies in humans, and more detailed animal studies, we hypothesize that ionizing radiation will lead to reduced parotid gland function and diminished salivary parenchymal tissue (with a preferential loss in acinar versus ductal cells). Further, we hypothesize that the parenchymal loss will increase with time (replaced by fat and connective tissue) and lead to progressive irreversible salivary dysfunction.

DETAILED DESCRIPTION:
Therapeutic irradiation to the head and neck for cancer damages salivary glands present in the radiation field. Despite long recognition of radiation-induced salivary hypofunction, and the associated oral morbidities, the specific damage mechanism(s) is not known and the structure and functional integrity of the surviving parenchymal tissue has not been well-documented. Detailed knowledge of the latter is particularly necessary in order to design appropriate corrective therapies. It is the purpose of this study to provide such a detailed structural and functional assessment of human parotid glands following irradiation. The study will examine 20 patients beginning just prior to therapeutic irradiation and continuing at intervals for 3 years for a total of 5 study visits. Study visits (prior to irradiation and at 4 weeks, 12 weeks, 12 months and 36 months post-irradiation) will include the following procedures: i) detailed oral exam and structured interview; ii) salivary gland functional assessment; iii) sialography of each parotid gland; iv) 99mTcO4 scan of the salivary glands; and v) a magnetic resonance imaging (MRI) scan of the parotid glands. Based on previous single observation studies in humans, and more detailed animal studies, we hypothesize that ionizing radiation will lead to reduced parotid gland function and diminished salivary parenchymal tissue (with a preferential loss in acinar versus ductal cells). Further, we hypothesize that the parenchymal loss will increase with time (replaced by fat and connective tissue) and lead to progressive irreversible salivary dysfunction.

ELIGIBILITY:
Age 21-80.

Diagnosis of head and neck cancer.

No surgery OR surgery with parotid glands intact.

Therapeutic radiation greater than or equal to 52 Gy.

Ambulatory.

No OR limited chemotherapy.

No Metastasis.

No allergy to Iodine.

No allergy to shellfish.

No metallic implants in head or neck.

No history of bleeding disorder.

No previous history of dry mouth (xerostomia).

No history of Sjogren's syndrome.

Negative HIV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1996-05; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States